CLINICAL TRIAL: NCT04045483
Title: A Randomized Controlled Crossover Trial to Assess Efficacy of Virtual Reality Based Cognitive Training Program in Mild Cognitive Impairment
Brief Title: Virtual Reality Based Cognitive Training Program in Mild Cognitive Impairment
Acronym: VRMCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inha University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-04-029
Record Dates: First submitted 2019-07-26; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Mild Cognitive Impairment
Keywords: virtual reality
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: This study is a single-blind, randomized, controlled, two-period crossover trial.
Who Masked: Outcomes Assessor
Masking Description: Raters of efficacy measures are blind to the group of a participant.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR based cognitive training (Experimental): Participants perform the VR based cognitive training under the supervision of a research nurse or psychologist for 30 min per session, twice per week, over the 6-week intervention period.
  Interventions: Other: Virtual reality based cognitive training
- Usual care (No Intervention): Participants take some medication for risk factors and cognitive impairment and receive health advice as a usual care.

INTERVENTIONS:
Other: Virtual reality based cognitive training — The VR-based cognitive training consists of a three-dimensional simulation of home, a mart, bus stop, and street. It provides an integrative cognitive training experience where participants are required to accomplish some common ADL's in three frequently visited places: home, a supermarket, and bus stop.
  Arms: VR based cognitive training

SUMMARY:
This study evaluates efficacy and safety of virtual reality (VR)-based cognitive training program in amnestic mild cognitive impairment.

DETAILED DESCRIPTION:
This study is a single-blind, randomized, controlled, two-period crossover trial. The intervention is done twice a week for 6 weeks. There are two arms. During the first period, participants were randomized to receive either VR-based cognitive training or usual care. After a 2-week washout period, the groups were crossed over to receive the alternative treatment for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50-85
2. A memory complaint by a participant or caregiver
3. Objective memory decline as defined by a delayed recall score of verbal learning test or logical memory worse than 1.0 standard deviations (SD) below age and education-adjusted normative mean
4. MMSE score better than1.5 SD below age and education-adjusted normative means
5. Global Clinical Dementia Rating (CDR) scale of 0.5 and memory score of CDR 0.5 or 1
6. Preserved activities of daily living (ADL), as defined by Korean Instrumental Activities of Daily Living < 0.4
7. Not demented
8. Hachinski Ischemic Score ≤ 4
9. Can read and write Korean
10. brain MRI or CT showing no other diseases capable of producing cognitive impairment
11. Having a reliable informant who could provide investigators with the requested information.
12. Provide written informed consent

Exclusion Criteria:

1. Participated in another clinical trial within the past 4 weeks
2. Other serious or unstable medical disease such as acute or severe asthma, severe or unstable cardiovascular disease, active gastric ulcer, severe liver disease, or severe renal disease
3. A clinically significant laboratory abnormality, such as an abnormal thyroid function test, abnormal low levels of vitamin B12 or folate, and positive syphilis serology
4. A primary other neurodegenerative disorder
5. Major psychiatric illness such as major depressive disorders
6. Drug or alcohol addiction during the past 10 years
7. Severe loss of vision, hearing, or communicative disability
8. Malignancy within 5 years
9. Any conditions preventing cooperation as judged by the study physician

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-07 (Actual); Primary Completion 2020-02-28 (Estimated); Study Completion 2020-03-14 (Estimated)

PRIMARY OUTCOMES:
Change of Short form of Literacy Independent Cognitive Assessment from baseline at 6 weeks | 6 weeks
  Measurement of memory, visuospatial function, language, and executive function The range of score is from 0 to 100. The higher score means better cognition.

SECONDARY OUTCOMES:
Change of Mini-Mental State Examination from baseline at 6 weeks | 6 weeks
  Evaluation of global cognition The range of score is from 0 to 30. The higher score means better cognition.
Change of Clinical Dementia Rating Scale-Sum of Boxes from baseline at 6 weeks | 6 weeks
  Evaluation of global cognition The range of score is from 0 to 18. The higher score means better cognition.
Change of Quality of life-Alzheimer's disease from baseline at 6 weeks | 6 weeks
  Evaluation of quality of life The range of score is from 0 to 52. The higher score means better quality of life.
Change of Geriatric Depression Scale-15 items from baseline at 6 weeks | 6 weeks
  Evaluation of mood The range of score is from 0 to 15. A higher score means more depression.
Change of Prospective and Retrospective Memory Questionnaire from baseline at 6 weeks | 6 weeks
  Evaluation of subjective memory The range of score is from 16 to 80. The higher score means more memory impairment.
Change of Bayer Activities of Daily Living from baseline at 6 weeks | 6 weeks
  Evaluation of activities of daily living The range of score is from 1 to 10. The higher score means worse ADL.

CONTACTS AND LOCATIONS:
Overall Officials: Seong Hye Choi, MD, PhD, Principal Investigator — Inha University Hospital
Locations (2):
- South Korea (2):
  - Inha University Hospital, Incheon
  - Ewha Womans University Mokdong Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No
We will decide it later.